CLINICAL TRIAL: NCT00117650
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Dose-Selection Study of Ad2/Hypoxia Inducible Factor (HIF)-1α/VP16 in Patients With Intermittent Claudication
Brief Title: Safety and Efficacy Study of Ad2/Hypoxia Inducible Factor (HIF)-1α/VP16 Gene Transfer in Patients With Intermittent Claudication
Acronym: WALK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PADHIF00704; 2004-002508-13 (EudraCT Number)
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease; Atherosclerosis
Keywords: leg pain; gene transfer; angiogenesis; Phase 2; Genzyme; peripheral arterial disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Atherosclerosis; Peripheral Arterial Disease | interventions — Hypoxia-Inducible Factor 1, alpha Subunit; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose (Active Comparator): 2 x 10^9 vp (viral particles)
  Interventions: Biological: Ad2/HIF-1α/VP16
- Middle Dose (Active Comparator): 2 x 10^10 vp
  Interventions: Biological: Ad2/HIF-1α/VP16
- High Dose (Active Comparator): 2 x 10^11 vp
  Interventions: Biological: Ad2/HIF-1α/VP16
- Placebo (Placebo Comparator): (PBS + 10% sucrose + 0.02% polysorbate 80)
  Interventions: Other: Saline (Placebo Control)

INTERVENTIONS:
Biological: Ad2/HIF-1α/VP16 — a one time treatment of 20 IM injections of 0.01 ML each into each leg for a total of 40 injections
  Other Names: HIF-1alpha
  Arms: Low Dose
Biological: Ad2/HIF-1α/VP16 — one time treatment of 20 IM injections of 0.01 ML each into each leg for a total of 40 injections.
  Other Names: HIF-1alpha
  Arms: Middle Dose
Biological: Ad2/HIF-1α/VP16 — a one time treatment of 20 IM injections of 0.01 ML each into each leg for a total of 40 injections.
  Other Names: HIF-1alpha
  Arms: High Dose
Other: Saline (Placebo Control) — a one time treatment of 20 IM injections of 0.01 ML each into each leg for a total of 40 injections.
  Arms: Placebo

SUMMARY:
The purpose of this Phase 2 clinical research study is to examine the safety of an experimental gene transfer agent, Ad2/HIF-1α/VP16, and its ability to stimulate the growth of new blood vessels from existing blood vessels (a process called angiogenesis) in an attempt to improve the flow of blood in the legs of patients with peripheral arterial disease (PAD).

Specifically, this study will enroll patients with severe intermittent claudication (IC) which is the stage of PAD in which a patient's walking ability is severely limited, causing pain in the legs upon exercise due to inadequate blood flow to the muscles of the lower limbs.

DETAILED DESCRIPTION:
This Phase 2 gene transfer study will look at whether different doses of Ad2/HIF-1α/VP16 can be tolerated safely by direct injection into the leg muscles where the blood flow is not sufficient to meet the oxygen demands of the leg muscles. The study will also assess whether patients who receive the investigational drug product are able to increase their maximal walking time using a standardized treadmill walking test.

The study design is a randomized, double-blind, placebo-controlled, parallel group, multi-center, Phase 2 dose-selection study. Seventy-five patients will be enrolled into each of 4 study drug groups (3 groups of Ad2/HIF-1α/VP16 gene transfer and 1 placebo group) for a total of 300 patients overall. Three different doses of Ad2/HIF-1α/VP16 gene transfer will be studied. The dose range was previously tested in animals and in the Phase 1 human studies. A placebo group is included in the study to compare safety and efficacy of different doses of Ad2/HIF-1α/VP16 with placebo. Each patient will receive a single set of 20 injections (100 μL each) of gene transfer or placebo in one administration to each leg for a total of 40 injections.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 40 to 80 years of age, inclusive.
* Clinical diagnosis of PAD, secondary to atherosclerosis, in both lower limbs, confirmed by objective evidence: An ankle-brachial index (ABI) of ≤ 0.90 at rest in at least 1 lower limb (Note: The index limb must be ≤ 0.90 at rest.); The ABI after exercise must be reduced by ≥ 20% from the ABI at rest in the index leg (the most symptomatic leg during the treadmill testing). The post-exercise ABI will also be performed on the other leg if the resting ABI > 0.90. A patient may be eligible for the study with a resting ABI in the non-index limb > 0.90 if: a. The post-exercise ABI in the non-index leg is also reduced by greater than or equal to 20% OR; b. A medically significant stenosis (defined as ≥ 50%) of a femoropopliteal or infrapopliteal artery is present, as documented via an imaging study (such as MR, conventional angiography, duplex ultrasound, or CT); If the ABI cannot be measured in either leg (due to non-compressible arteries), then a toe-brachial index (TBI) of ≤ 0.70 may be used in its place to confirm PAD.
* Symptoms of severe intermittent claudication (IC) in at least 1 lower limb persisting for ≥ 6 months
* Patients with a peak walking time (PWT) of 1 to 12 minutes (inclusive) using the standardized exercise treadmill test at each of the 2 consecutive treadmill tests performed at least a week apart during the Screening period.
* During Screening, patients must demonstrate consistency of PWTs between 2 standardized exercise treadmill tests (Walk 1 and Walk 2) performed at least 1 week apart.
* Consistency of the PWT between the 2 visits is achieved if the difference between PWT at Walk 1 and Walk 2 is ≤ 25% of the higher of the 2 PWTs ([higher PWT - lower PWT]/higher PWT).
* If the difference between PWT at Walk 1 and Walk 2 is > 25% of the higher of the 2 PWTs, a third treadmill test (Walk 3) may be performed at the discretion of the Principal Investigator between 7 and 14 days following Walk 2. The variability in PWT warranting the performance of Walk 3 must be secondary to circumstances that may contribute to the observed variation (e.g., prior exertion, inconsistent timing, ingestion of a meal within 4 hours, etc). To qualify for the study, the difference between PWT of either Walk 1 or Walk 2 as compared with Walk 3 must be ≤ 25% of the higher of the 2 PWTs ([higher PWT - lower PWT]/higher PWT). The decision whether Walk 1 or Walk 2 will be used for comparison with Walk 3 will be made prospectively and reviewed with the Sponsor.
* An acceptable mean PWT must be achieved within 4 weeks of treatment administration.
* Patients have been considered for other potential treatment options including exercise rehabilitation, smoking cessation, and pharmacological therapy prior to Enrollment.
* Claudication severity, concomitant medications for the treatment of CAD, PAD, and IC, smoking status and exercise habits should be clinically stable for 3 months prior to Enrollment.
* Patients who are committed to following the protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

* Patients with either current or any history of Critical Limb Ischemia (CLI; that is, patients classified as Rutherford Category 4 [ischemic rest pain], Rutherford Category 5 [non-healing ischemic ulcers and minor tissue loss], or Rutherford Category 6 [non-healing ischemic ulcers and major tissue loss]).
* Patients in whom arterial insufficiency in the lower extremity is the result of acute limb ischemia or an immunological or inflammatory non-atherosclerotic disorder (eg, thromboangiitis obliterans [Buerger's Disease]) and systemic sclerosis [both limited and diffuse forms]).
* A PAD-specific surgical revascularization procedure within 6 months of enrollment or a PAD-specific percutaneous procedure within 3 months of enrollment, or patients likely to require a PAD-specific revascularization procedure within 6 months after Enrollment.
* Patients with aortoiliac disease that limits inflow in either leg: a. Patients with concomitant aortoiliac disease (i.e., patients with a significant component of inflow disease in the distal aorta, common or external iliac, or proximal common femoral artery) as assessed by an imaging modality (e.g., segmental limb pressures and waveform analysis, duplex ultrasound scanning, magnetic resonance angiography, or radio-contrast arteriogram) performed within 1 year prior to Enrollment. If subject has had a bypass after the imaging study, then documentation of graft patency is required within 6 months prior to Enrollment; b. If it is suspected at Screening that a patient has aortoiliac disease based on vascular examination, an imaging modality (e.g., segmental limb pressures and waveform analysis, duplex ultrasound scanning, magnetic resonance angiography, or radio-contrast arteriogram) must be performed to rule it out if there is not one available within the times specified above. If there is no suspicion of aortoiliac disease in the Principal Investigator's judgment, an imaging test at Screening is not required for study purposes.
* Patients in whom walking impairment due to pain in the index leg is the result of these nonatherosclerotic comorbid conditions: venous claudication, chronic compartment syndrome, peripheral nerve pain (e.g., severe peripheral neuropathy), pseudoclaudication caused by spinal cord compression, or acute limb ischemia which, in the Principal Investigator's judgment are severe enough to confound the assessment of the patient's IC.
* Conditions other than IC of significant severity that could confound PWT on the standardized exercise treadmill test causing premature or inconsistent termination of exercise (e.g., angina pectoris, heart failure [New York Heart Association {NYHA} Classes III and IV], respiratory disease [e.g., chronic obstructive pulmonary disease], orthopedic disease, neurological disorders, rheumatologic disorders [e.g., severe degenerative joint diseases], dyspnea, fatigue, prior lower limb amputation, including amputations proximal to the metatarsal or phalangeal joints).
* Presence or history of cancer within 5 years of enrollment or not current with recommended screening guidelines for colorectal, lung, prostate, breast, cervical, and uterine cancers, with the exception of low grade and fully resolved non-melanoma skin malignancy.
* Patients with a well-defined clinical or genetic disorder predisposing to malignancy should be excluded (e.g., von Hippel Lindau, familial polyposis coli, BRCA1, BRCA2, etc).
* Patients with baseline funduscopic evidence of active proliferative diabetic retinopathy, preproliferative diabetic retinopathy, or wet AMD AND/OR Patients with a history of treatment for active proliferative diabetic retinopathy or wet AMD within 5 years of enrollment.
* Diabetes type 1 (juvenile onset)
* Poorly controlled type 2 diabetes (ie, HbA1C >10%) at Screening
* Active hepatitis defined as clinically significant increase in liver enzymes (ie, 3 times the ULN) or other current infectious disease
* Patients with symptoms of respiratory infection at time of Screening and/or randomization period and/or patients who have been on systemic or oral antibiotics for active infection within 2 weeks of study drug administration.
* Patients with clinically significant abnormal hematology (eg, hematocrit < 30%, white blood cell count > 14,000), blood chemistry, renal, hepatic, or other laboratory parameters that could be the result of an underlying malignancy or systemic infection (e.g., serum creatinine ≥ 2.5 mg/dL), as judged by the investigator.
* Patients with the following comorbidities who may not be healthy enough to successfully complete all protocol requirements or in whom results may be particularly difficult to assess: Concurrent severe congestive heart failure (NYHA Classes III and IV); Life-threatening ventricular arrhythmias, unstable angina (characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged duration), and/or myocardial infarction within 4 weeks before enrollment; Coronary artery bypass grafting or percutaneous coronary intervention within 3 months before enrollment; A renal and/or carotid revascularization procedure within 1 month of enrollment; Transient ischemic attack within 3 months before enrollment; Deep vein thrombosis within 3 months before enrollment; Severe chronic obstructive pulmonary disease (room air arterial PO2 < 60 mmHg or PCO2 > 50 mmHg, or abnormal pulmonary function tests (FEV1 < 1.2 L/sec); Thrombocytopenia (defined as platelet count < 100,000/mm3); Undergoing hemodialysis; Patients with immunocompromised conditions, organ transplant recipients and/or need for immunosuppressive therapy; Neurological dementia (i.e., Alzheimer's Disease); Hemorrhagic stroke
* Patients with a known allergy to the vehicle, placebo control, or any other medications or imaging agents required for participation in this study.
* Fertile women who are pregnant (as confirmed by a serum pregnancy test at the Screening Visit and a urine pregnancy test at Day 0 prior to study drug administration), nursing, or using either no or an inadequate form of contraception.
* Fertile men and women who are not willing to use barrier-type contraception for at least 90 days post-treatment.
* Patients with a recent history of alcoholism or drug abuse, or severe emotional, behavioral or psychiatric problems, who may not be able to adequately comply with the requirements of the study.
* Patients receiving experimental medications or participating in another study using an experimental drug or experimental procedure within 30 days of enrollment into this study.
* Patients previously enrolled in a prior angiogenic gene therapy clinical study, unless patient was a known placebo patient.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Peak Walking Time | at 6 months

SECONDARY OUTCOMES:
Peak walking time | at 3 months and at 1 year
Claudication onset time | at 3 months, 6 months, and at 1 year
Quality of life questionnaires | at 3 months, 6 months, 1 year
Resting ankle brachial index | at 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (47):
- United States (35):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California at Davis, Sacramento, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - The Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Heart Institute, Atlantis, Florida
  - Baptist Health Care, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois
  - The Care Group at the Heart Center, Indianapolis, Indiana
  - Ochsner Clinic Foundation, Metairie, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, CCP4C, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
- Germany (6):
  - Ev. Krankenhaus Königin Elisabeth, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Klinikum Karlsbad Langensteinbach gGmbH, Karlsbad
  - Universitätsklinikum Schleswig Holstein/Campus Luebeck, Lübeck
  - Klinikum Grosshadern, Munich
  - Universitätsklinikum Munster, Münster
- United Kingdom (6):
  - Belfast City Hospital, Belfast
  - Selly Oak Hospital, Birmingham
  - Ninewells Hospital & Medical School, Dundee
  - Hull Royal Infirmary, Hull
  - St. George's Hospital and Medical School, London
  - Ealing Hospital, Southall, Middlesex

REFERENCES:
- [Derived] Creager MA, Olin JW, Belch JJ, Moneta GL, Henry TD, Rajagopalan S, Annex BH, Hiatt WR. Effect of hypoxia-inducible factor-1alpha gene therapy on walking performance in patients with intermittent claudication. Circulation. 2011 Oct 18;124(16):1765-73. doi: 10.1161/CIRCULATIONAHA.110.009407. Epub 2011 Sep 26. PMID 21947297